CLINICAL TRIAL: NCT00999323
Title: Endothelial Function and Heart Rate Variability After Stenting in Coronary Arteries
Brief Title: Endothelial Function and Heart Rate Variability After Stenting
Acronym: FUNKIS
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2007.061.07
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2009-10

CONDITIONS: Restenosis or Adverse Cardiovascular Event

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma and full blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary artery disease: patients who have been revascularized by PCI with stent implantation due to an acute coronary syndrome
  Interventions: Device: stent implantation in coronary artery

INTERVENTIONS:
Device: stent implantation in coronary artery — Percuatenous Coronary Intervention with implanatation of a stent

SUMMARY:
The objective of this study is to evaluate whether impaired endothelial function and low heart rate variability are associated with clinical restenosis after percutaneous coronary intervention with stent implantation in patients with angina or acute coronary syndrome.

Furthermore, the study examines a potential correlation between biomarkers of endothelial cell activation and endothelial dysfunction.

DETAILED DESCRIPTION:
Background Atherosclerosis is a chronic, systemic and diffusely distributed disease causing focal complications in different vascular beds.

Impaired endothelial function is the initial step in the progressive course of atherosclerosis . Endothelial dysfunction is considered a systemic process and both coronary and peripheral endothelial dysfunction have been shown to be independently associated with cardiovascular events .

Percutanenous coronary intervention (PCI) with implantation of stent is the treatment of choice in symptomatic stenotic coronary artyery disease (CAD), but in-stent restenosis and progression of disease remains its main limitation. Early identification of patients at risk of restenosis after PCI would therefore be of clinical value. There is only limited prospective data on the role of peripheral endothelial dysfunction after PCI predicting restenosis and cardiovascular events , , .

Furthermore, it is unknown if peripheral endothelial dysfunction is associated with increased levels of biomarkers of endothelial cell activation in this population.

There are conflicting data on inflammatory markers as high-sensitivity CRP with regard to endothelial function.

Low heart rate variability (HRV) predicts automic dysfunction and is a strong and independent predictor of mortality in patients with coronary artery disease (CAD) . Clinical depression after myocardial infarction is associated with decreased HRV, linking depression to increased cardiac mortality in post-myocardial infarction patients . Whether decreased HRV is associated with endothelial dysfunction or restenosis is unknown.

Objective The objective of this study is to evaluate whether impaired endothelial function and low HRV are associated with clinical restenosis.

Furthermore, the study examines a potential correlation between biomarkers of endothelial cell activation and endothelial dysfunction.

Another issue is depression after PCI and a potential association with impaired endothelial function and increased levels of makers for endothelial activation.

Methods

Subjects This prospective study includes consecutively patients with acute coronary syndromes undergoing PCI with stent implantation for significant single vessel disease at Stavanger University Hospital, Stavanger, Norway. Patients will be followed for at least 6 months.

Exclusion criteria are multivessel disease, left ventricular dysfunction defined as ejection fraction (EF) < 50%, former aortocoronary bypass-surgery, systemic inflammatory diseases other than atherosclerosis, cognitive impairement, severe psychiatric disorder, renal failure (kreatinin > 250 mmol/l), refusion to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients after successful revascularization by percutaneous coronary intervention with stent implantation for single coronary artery disease

Exclusion Criteria:

* Multivessel coronary artery disease
* Left ventricular dysfunction defined as ejection fraction (EF) < 50%
* Former aortocoronary bypass-surgery
* Systemic inflammatory diseases other than atherosclerosis
* inability to give informed consent
* Renal failure (kreatinin > 250 mmol/l)
* Refusion to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who have been revascularized by coronary intervention with stent implantation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
clinical restenosis, major cardiovascular event | 12 months

SECONDARY OUTCOMES:
endothelial function, heart rate variability | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stavanger University Hospital, Stavanger, Norway